CLINICAL TRIAL: NCT04961437
Title: Evaluation of Dyspnea, Pulmonary VentIlation and DIaphragmatic Function in de Novo Adult Acute Respiratory Failure.
Brief Title: Impact of Dyspnea, Regional Lung Ventilation, and Diaphragmatic Function During de Novo Acute Respiratory Failure
Acronym: DY-VI-DI
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00329-32
Record Dates: First submitted 2021-06-18; First posted 2021-07-14 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Acute Respiratory Failure
Keywords: Acute respiratory failure; diaphragm; dyspnea; EIT
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with de novo acute respiratory failure: The following tests will be performed as part of the research (these tests are usually performed as part of routine care but not routinely and comprehensively):
  * A diaphragmatic ultrasound in the half-seated position. Diaphragmatic excursion and thickening fraction will be measured in the right hemi-diaphragm.
  * A 10-minute reference acquisition. They will be performed at inclusion, H2, H4 and H48.
  Interventions: Other: Diaphragmatic ultrasound and electrical impedance tomography

INTERVENTIONS:
Other: Diaphragmatic ultrasound and electrical impedance tomography — A diaphragmatic ultrasound in a half sitting position. The diaphragmatic excursion and the thickening fraction of the right hemi-diaphragm will be measured.
  - Acquisition of 10 minutes of regional pulmonary ventilation by electrical impedance tomography.

SUMMARY:
Modern management of acute respiratory failure aims to relieve dyspnea and anxiety by providing a non-invasive respiratory support. This approach tries to avoid endotracheal intubation, patient self inflicted lung injuries (PSILI) and diaphragmatic dysfunction. The present study aims to evaluate dyspnea, pulmonary regional ventilation and diaphragmatic function in patients with hypoxemic acute respiratory failure by different observations, and to bring risk factor for intubation out.

DETAILED DESCRIPTION:
Patients aged of 18 years or more, presenting with an acute respiratory failure without hypercapnia will be included in the study. Clinical and biological variables, dyspnea assessment, regional lung ventilation (electrical impedance tomography) and diaphragm function (ultrasound) will be evaluated at inclusion and at 2 hours, 4 hours and 48 hours after inclusion. In case of intubation, diaphragmatic function will be also evaluated with phrenic nerve stimulation technique.

Primary endpoint is intubation at day 7. Secondary endpoints are measurement of dyspnea, pulmonary ventilation and diaphragmatic function, also ventilator free days, ICU length of stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Acute respiratory insufficiency defined by the three following items :

  1. PaO2/ FiO2 <300
  2. Respiratory rate > 25/min
  3. Oxygen support > 10L/min or High Flow nasal oxygen (HFNO)
* Non opposition by the patient to be included
* Social insurance

Exclusion Criteria:

* Respiratory acidosis (pH < 7,35 PaCO2 > 45mmHg or 6kPa)
* Chronic respiratory disease ( COPD, bronchiectasis…)
* Cardiogenic Acute lung oedema
* Non intubation decision at randomisation
* Contraindication for Electro-impedance tomography-belt placement (chest trauma with rib fractures, thoracic wound, chest tube).
* Uncommunicative patient (Glasgow coma scale <12)
* Guardianship or curators for vulnerable patients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with de novo acute respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
Oro-tracheal intubation | 7 days after admission in the ICU
  Patients who will be intubated within the 7 days after admission in the ICU

SECONDARY OUTCOMES:
Diaphragmatic function | 2 days after inclusion
  using ultrasonography, measure of diaphragmatic excursion and diaphragmatic thickening in Hertz (Hz)
Diaphragmatic function | 2 days after inclusion
  Diaphragmatic function evaluation by phrenic nerve stimulation (only for intubated patients).
lung regional ventilation | 2 days after inclusion
  As measured with Electric Impedance Tomography index measures (inhomogeneity index, end expiratory lung impedance change)
Dyspnea evaluation | 28 days after inclusion
  Dyspnea evaluation using visual analogue scale applied to dyspnea: from 1 to 10, 1 corresponding to "no breathlessness" and 10 to "maximum breathlessness".
Dyspnea evaluation | 28 days after inclusion
  Dyspnea evaluation using Respiratory Distress Observation Scale (RDOS)
Mechanical ventilation duration | 28 days after inclusion
  (only for intubated patients).
ICU length of stay | 28 days after inclusion
  for all patients
ICU mortality | 28 days after inclusion
  for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Martin DRES, MD PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière", Intensive care unit, Paris, France

IPD SHARING:
Plan to Share IPD: No